CLINICAL TRIAL: NCT05004493
Title: Assessment of Changes in Normal and Pathological Immune Factors in Patients Undergoing Plasma Exchange
Brief Title: Biorepository and Registry for Plasma Exchange Patients
Status: Recruiting | Type: Observational
Sponsor: Charles M Knudson (Other)
Responsible Party: Sponsor-Investigator, Charles M Knudson, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202104462
Record Dates: First submitted 2021-08-05; First posted 2021-08-13 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Antibody-mediated Rejection; NMO Spectrum Disorder; TTP; CIDP
Keywords: plasma exchange; plasmapheresis
MeSH Terms: conditions — Neuromyelitis Optica; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Plasma samples collected during and after the course of plasma exchange treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Plasma arm: Patients receiving plasma as one of the main replacement fluids
- No Plasma: Patients receiving saline and/or 5% albumin as the replacement fluid.

SUMMARY:
Patients who have immune mediated diseases commonly undergo plasma exchange (PLEX) procedures to remove pathological substances, typically believed to be antibodies. At our facility about 400 of these procedures are performed annually on 40-60 different patients. These procedures are considered within the standard of care for these patients and are covered by insurance. This study will not influence the treatment plan for subjects who participate in this study. The goal of the study is to collect and cryopreserve blood biospecimens (plasma, serum, PBMCs) for current and future studies. Any patient undergoing plasma exchange procedures will be eligible for the study. Patients or the legally authorized representative (LAR) will be consented for the study as soon as feasible after the are referred to DeGowin for plasma exchange. The immediate objective of the study is to examine antibody levels (IgG/IgM) and BAFF levels in the blood of these patients over the course of the plasma exchange treatments. Specimens and clinical data will be collected such that other immune factors that may regulate B cell survival, proliferation and antibody secretion can be studied. Another goal of the study is to isolate and cryopreserve PBMCs at different points during the patient's treatment. This would allow the study of immune cells that may mediate these diseases. The study will also follow pathological antibodies over time in these patients so biospecimens can be obtained even after the completion of their course of plasma exchange treatments. The collection of biospecimens and clinical information from these subjects will help us understand the impact of plasma exchange on both normal and pathological immune factors in a variety of patients undergoing these procedures.

ELIGIBILITY:
Pts undergoing plasma exchange therapy are eligible to be in this protocol

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients > 12 years old who are undergoing plasma exchange therapy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
IgG and IgM antibody levels | Levels over the course of treatment will be compared. Typically 1-2 weeks.
  The effect of replacement fluids on IgG and IgM antibody levels will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- DeGowin blood Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data may be shared with other investigators on a case by case basis.

REFERENCES:
- [Background] Winters JL. Plasma exchange: concepts, mechanisms, and an overview of the American Society for Apheresis guidelines. Hematology Am Soc Hematol Educ Program. 2012;2012:7-12. doi: 10.1182/asheducation-2012.1.7. PMID 23233554
- [Background] Reeves HM, Winters JL. The mechanisms of action of plasma exchange. Br J Haematol. 2014 Feb;164(3):342-51. doi: 10.1111/bjh.12629. Epub 2013 Oct 30. PMID 24172059
- [Background] Mockel T, Basta F, Weinmann-Menke J, Schwarting A. B cell activating factor (BAFF): Structure, functions, autoimmunity and clinical implications in Systemic Lupus Erythematosus (SLE). Autoimmun Rev. 2021 Feb;20(2):102736. doi: 10.1016/j.autrev.2020.102736. Epub 2020 Dec 14. PMID 33333233
- [Background] Schiemann B, Gommerman JL, Vora K, Cachero TG, Shulga-Morskaya S, Dobles M, Frew E, Scott ML. An essential role for BAFF in the normal development of B cells through a BCMA-independent pathway. Science. 2001 Sep 14;293(5537):2111-4. doi: 10.1126/science.1061964. Epub 2001 Aug 16. PMID 11509691